CLINICAL TRIAL: NCT02121886
Title: To Evaluate the Safety and Outcome of the Parietal Peritoneum as a Substitute Graft for Venous Reconstruction in Hepatobiliary and Pancreatic Surgery
Brief Title: The Parietal Peritoneum as a Substitute Graft for Venous Reconstruction in HPB Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beaujon Hospital (Other)
Responsible Party: Principal Investigator, Safi Dokmak, MD, Beaujon Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Departement of HPB surgery; Departement of HPB surgery (Other: Beaujon Hospital, Clichy, France)
Record Dates: First submitted 2014-04-20; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Safety; Availability; Venous Patency; Oncological Benefits; Morbidity
MeSH Terms: interventions — Hepatectomy; Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parietal peritoneum (Experimental)
  Interventions: Procedure: venous reconstruction with the parietal peritoneum

INTERVENTIONS:
Procedure: venous reconstruction with the parietal peritoneum
  Other Names: Liver resection; Pancreatic resection; Venous resection; Reconstruction; Parietal peritoneum

SUMMARY:
To evaluate the safety and outcome of the parietal peritoneum for venous reconstruction HPB surgery. Although the parietal peritoneum had already been used and published for the reconstruction of the vena cava, however this one was never described or described in HPB surgery

DETAILED DESCRIPTION:
Improvements in surgical techniques, perioperative management and effective chemotherapy regimens, have increased the resectability of malignant hepatobiliary and pancreatic tumors when associated with vascular invasion. Therefore, simultaneous vascular resection is increasingly required to obtain an adequate resection margin and improve patient definite survival. Although most vascular resection associated with pancreatectomy can be reconstructed by simple venorraphy or end-to-end anastomosis, a segmental or lateral vacular graft (VG) can be necessary in 8-12 % of cases. Vascular reconstruction can be planned preoperatively if the vascular invasion is evident and an appropriate VG can be prepared. Differents sources of VG are available including autogenous veins , synthetic such as polytetrafluoroethylene (PTFE) , cryopreserved and veins from the resected liver. However the decision to perform vascular resection may be made during dissection due to vascular invasion or injury and even occasionnally taken while the mesentericoportal vein (MPV) or vena cava (VC) are occluded. In this emergency situation, an urgent and easily available graft is necessary to prevent prolonged ischemia. The difficulty of anticipating the need for these vascular resections during HPB surgery, has lead certain authors including those in our group to use either the veins from the resected liver, the umbilical vein or the parietal peritoneum (PP) for vena cava reconstruction. The aim of our study is to evaluate the safety and outcome of the parietal peritoneum as a substitute patch for venous reconstruction during HPB surgery in emergency and elective situations.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to HPB unit and schudeled for major liver or pancreatic resections with suspected venous invasion. Venous invasion is suspected on CT scan (vein narrowing or disappearance of the fat plane between the vein and the tumor) performed within 1 month of surgical resection. Informed consent will be obtained and the parietal peritoneum will be used as a substitute graft for resection-reconstruction in these patients if intra-operative exploration confirmed this venous invasion

Exclusion Criteria:

* Patients who refuse to participate and patients with suspected peritoneal carcinomatosis or if intra-operative exploration confirmed the presence of peritoneal carcinomatosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Safety and venous patency | Up to 4 months
  The primary outcome of this study will be the safety and venous patency. Safety means "to see if the parietal peritoneum is rigid and there is no tearing of bleeding in the reconstructed area, related to venous pressure", this safety will be assessed clinically (exteriorized bleeding from the reconstructed zone and on CT scan to search for local hematoma). Patency will be assessed by regular CT scan performed on postoperative day 8,30,90 and 120. On CT scan, this evaluation will include the degree on venous stenosis (0%, <25%, 25%-75%, >75%, thrombosis) compared to non reconstructed vein, the presence of thrombosis with collateral venous circulation or venous enlargement in the reconstructed area

SECONDARY OUTCOMES:
Long-term venous Patency | Up to 6 months
  The venous latency will be assessed at 6 months of the surgical resection and the assessment with be done by CT scan in order to study the degree of venous stenosis, the presence or not of thrombosis or collateral venous circulation and venous enlargement.

OTHER OUTCOMES:
Oncological benefit and rate or R0 venous resection | up to 1 month
  We will study on histology the rate of R0 resection (margins tumor free) in order to see if this technique allow us to resect largely the tumor with the benefit to increase the rate of R0 resection on the vein and surrounding structures

CONTACTS AND LOCATIONS:
Locations (1):
- Departement HPB surgery, Beaujon Hospital, Clichy, Hauts de seine, France

REFERENCES:
- [Derived] Dokmak S, Aussilhou B, Sauvanet A, Nagarajan G, Farges O, Belghiti J. Parietal Peritoneum as an Autologous Substitute for Venous Reconstruction in Hepatopancreatobiliary Surgery. Ann Surg. 2015 Aug;262(2):366-71. doi: 10.1097/SLA.0000000000000959. PMID 25243564